CLINICAL TRIAL: NCT06826235
Title: Tip 2 Diyabetli Yetişkin Bireylerde Hurma Tüketiminin Hedonik Açlık ve İştah Hormonları Üzerine Etkilerinin İncelenmesi
Brief Title: Investigation of the Effect of Date Consumption on Hedonic Hunger and Appetite in Adult Individuals With Type 2 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, AYŞE ÇAMLİ, Research Assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 06.03.2024-26185
Record Dates: First submitted 2025-01-23; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Type 2 Diabetes Mellitus; Appetite
Keywords: date; hedonic hunger; appetite; type 2 diabetes; lipid profile
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: control and intervention group
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INTERVENTION GROUP (Experimental)
  Interventions: Other: 3 dates at the breakfast meal in the diet program
- CONTROL GROUP (No Intervention)

INTERVENTIONS:
Other: 3 dates at the breakfast meal in the diet program — Participants in the intervention group will consume 3 dates at the breakfast meal in the diet program.
  Arms: INTERVENTION GROUP

SUMMARY:
The aim of this study was to investigate the effects of date consumption on hedonic hunger and appetite hormones in individuals diagnosed with type 2 diabetes.The main questions it aims to answer are:

* Does date consumption reduce hedonic hunger in individuals with type 2 diabetes?
* Does persimmon consumption change Ghrelin, GLP-1 and GIP concentrations in individuals with Type 2 diabetes?
* Does persimmon consumption reduce HOMA-IR and HbA1c values in individuals with Type 2 diabetes?
* Does consumption of persimmon reduce LDL cholesterol, total cholesterol and triglyceride concentrations in individuals with type 2 diabetes? To see the effects of date consumption on hedonic hunger and appetite hormones, the researchers will compare individuals with type 2 diabetes who consume 3 dates daily with individuals with type 2 diabetes who do not.

Participants:

* Individuals in the intervention group will consume 3 (25 g) Baghdad dates (15 g CHO) daily as part of the breakfast meal, while individuals in the control group will not consume dates.
* Three interviews will be conducted with patients.
* A record of blood findings and questionnaires will be kept during these interviews.

DETAILED DESCRIPTION:
1. Study Design and Participants The sample of this randomised controlled clinical trial will consist of adult individuals with Type 2 diabetes who apply to Erzurum City Hospital Internal Medicine outpatient clinic. A control group will be formed with individuals with Type 2 diabetes in the same age group. Informed Voluntary Consent Form will be obtained from the individuals before starting the study. Power analysis was performed to determine the sample size. The study population was determined as 70 individuals with the G-power programme. In this randomised controlled study, individuals will be randomly assigned to the intervention and control groups using a computer generated list.
2. Intervention and Control Groups Individuals who agree to participate in the study will be randomly assigned to the intervention and control groups. The study consists of three stages. The first interview will take place at week 0, the second interview at week 6 and the last interview at week 12. The control group will not be intervened by not giving any additional food and will be asked not to consume dates during the study. The intervention group will be informed at the first interview about which meal and in what quantity they will consume dates. Dates will be delivered to participants at baseline (6-week supply) and at week 6 of the study (6-week supply). Individuals in the intervention group will consume 3 (25 g) Baghdad dates (15 g CHO) daily as part of the breakfast meal. Individuals will be given weekly recording sheets to record their date consumption. The diaries will be collected fortnightly to ensure dates are consumed as directed (a photo of the diary will be requested via email or social media). Individuals will receive a fortnightly telephone reminder.
3. Questionnaire Form Information such as socio-demographic characteristics, smoking and alcohol consumption status, health status, medication used in diabetes treatment, etc. will be obtained through a face-to-face questionnaire. Visual Analogue Scale (VAS) will be used for subjective hunger. The questionnaire form will also include the Food Power Scale for the assessment of hedonic hunger, the International Physical Activity Questionnaire short form (IPAQ-SF) for the assessment of physical activity levels and three-day Food Consumption Records for the assessment of food consumption.
4. Anthropometric Measurements In the study, anthropometric measurements of individuals will be taken at 0. 6. and 12. weeks. Height will be measured with a stadiometer (SECA 213) with an accuracy of 0.1 cm with the feet side by side and the head in the Frankort plane. Bioelectrical impedance analysis (BIA) (TanitaBC-730) will be used to evaluate body weight and body composition. The measurements will be performed by the researcher.
5. Biochemical analyses Blood samples taken from the individuals at weeks 0 and 12 will be analysed in the Biochemistry Laboratory of Atatürk University Research Hospital. Fasting blood glucose, fasting blood insulin, HbA1c, Ghrelin, GLP-1, GIP total cholesterol, LDL cholesterol and triglyceride analyses will be performed. Fasting blood glucose, fasting blood insulin, HbA1c, total cholesterol, LDL cholesterol and triglycerides are the tests routinely requested by the doctor. Blood samples for ghrelin, GLP-1 and GIP analyses will be collected and analysed separately in the laboratory. Fasting blood glucose and insulin values of individuals who will be used in homeostatic model assessment for insulin resistance (HOMA-IR) will be measured. Fasting and postprandial blood glucose will be measured with a glucometer at 0, 6 and 12 weeks of the study.

   * Statistical analyses will be performed using SPSS version 22 software.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with Type 2 diabetes aged 19-50 years (excluding menopausal women),
* Individuals with BMI between 25-35 kg/m2,
* Individuals with a Nutritional Strength Scale score of 2.5 and above,
* Individuals who agreed not to start taking new dietary supplements or alternative therapies during the study period,
* Individuals who agree not to change their current physical activity level and diet.

Exclusion Criteria:

* Individuals who do not approve the volunteer consent form,
* Individuals with a Nutritional Strength Scale score below 2.5,
* Pregnant or breastfeeding women (or women planning to become pregnant within 3 months)
* Individuals with dietary energy <800 kcal/day and >4000 kcal/day,
* Individuals with pre-diabetes, type 1 diabetes and gestational diabetes,
* Individuals with HbA1c >10
* Individuals taking antibiotics or hormone replacement therapy History of malignancy (except non-melanoma skin cancer).
* Individuals with regular consumption of dates before inclusion in the study,
* Individuals diagnosed with Type 2 diabetes using insulin and oral antidiabetic drugs with thiazolidinedione active substance,
* Individuals with a history of diabetic ketoacidosis, diabetic coma or precoma within 6 months prior to the date of admission; serious infections, surgery, serious trauma requiring insulin treatment, haemodialysis treatment (including peritoneal haemodialysis), serious liver injury and serious vascular complications (stroke, myocardial infarction and heart failure) requiring hospitalisation,
* Individuals taking pharmacological agents that have effects on appetite such as psychotropics, antiepileptics, antidepressants, antipsychotics and/or steroids,
* Individuals diagnosed with eating disorders and/or psychological disorders,
* Individuals with physical illnesses that affect eating behaviour or appetite, such as uncontrolled hyperthyroidism or hypothyroidism, Cushing's disease, acromegaly, adrenal insufficiency, chronic renal failure (stage 4 or 5), tuberculosis, human immunodeficiency virus (HIV) infection.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-05-14 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Appetite hormone levels | 3 months
  GLP-1, GIP and Ghrelin hormone levels in plasma will be measured in pg/ml.
Hedonic hunger levels | 3 months
  Hedonic hunger levels of individuals will be determined using the Power of Food Scale (PFS).

CONTACTS AND LOCATIONS:
Locations (1):
- Erzurum City Hospital, Erzurum, Palandöken, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No